CLINICAL TRIAL: NCT03598361
Title: Evaluation of Mineral Status in Pregnant Women and Its Association With Fetal Development
Brief Title: Mineral Status in Pregnant Women
Acronym: PREDISH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Joanna Suliburska, Principial Investigator, Poznan University of Life Sciences
Other Study IDs: 297/17
Record Dates: First submitted 2018-07-01; First posted 2018-07-26 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Pregnancy; Disorder, Blood
Keywords: pregnancy outcomes, minerals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples hair amniotic fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ensuring an adequate supply of nutrients, which include trace elements, is particularly important in pregnancy. Both deficiency and excess of trace elements in the body can interfere with conception and maintaining a healthy pregnancy. The effects of malnutrition and shortages in fetal life may increase the risk of miscarriages, congenital malformations, premature births, intrauterine fetal growth restriction (IUGR) and more frequent perinatal mortality. Nutritional deficiencies during fetal development may also have long-term consequences for the child, such as disorders in his biological and psychomotor development.

In women of procreative age, an adequate supply of minerals, especially iron, calcium, zinc, magnesium and copper, is very important. The results of clinical trials indicate an association of anemia in pregnant women with premature delivery and low birth weight of a newborn. Calcium deficiency leads to the development of hypertension in pregnancy (including preeclampsia) and increases the risk of premature birth. Deficiency of zinc and copper in the mother's body is associated with complications of pregnancy and childbirth and affects inappropriate fetal development.

The deficiency of these mineral components is often observed in young women-potential mothers. Increasing during pregnancy the need for nutrients and abnormal nutrition, intensify the deficiencies of minerals and affect the abnormal development of the fetus. It seems that during the course of pregnancy, changes in the mineral nutrition of women can be observed, which is why it is important to monitor this condition in the subsequent months of pregnancy.

Due to the above, the aim of the planned research is to determine the nutrition and nutritional status of women in the subsequent trimesters of pregnancy.

Obtained results will allow to formulate appropriate nutritional recommendations and / or indicate the need to implement appropriate mineral supplementation for women in every trimester of pregnancy.

DETAILED DESCRIPTION:
Assumptions of the research, description of the study group (age, sex, health status, size of the group):

The review of literature on the subject shows that there are relationships between the concentrations of certain elements (especially magnesium, copper, cadmium and barium), and the gestational age and fetal biometric parameters. Scientific research carried out so far has also pointed to the relationship between pregnancy-related diseases (pre-eclampsia, intra-uterine growth disorders) and the mineral status of pregnant women. Little is known about the minerals concentration in amniotic fluid. The main aim of the study is to determine the correlation between the mineral status of pregnant women and the course of pregnancy and fetal development. During the tests, the concentrations of selected mineral components in the maternal blood serum, amniotic fluid and the hair of pregnant women will be determined. The obtained data will be combined with dietary data obtained through a questionnaire and nutrition journal. The dependence between the content of minerals in the analyzed material and the fetus development, the health of the newborn and the course of pregnancy will also be assessed. Clear identification of the correlation between the mineral status of pregnant women and the course of pregnancy and fetal development may be an important contribution to the development of science about nutrition during pregnancy and prenatal diagnosis and prevention of pregnancy complications.

The importance of research:

The review of the literature on the subject shows that there are few studies showing correlations between the concentration of minerals in various compartments of the pregnant woman's body, and the course of pregnancy and fetal development. There is also a lack of data on the relationship between diet and supplementation during pregnancy and the mineral status of pregnant women.

The planned studies are intended to determine the concentration of minerals, e.g. in materials such as blood serum, amniotic fluid, or hair. Elemental analysis of hair will allow assessment of long-term nutritional status of women with mineral components. The mineral composition of amniotic fluid, according to literature data, requires further analysis. It is suggested that amniotic fluid may be an important diagnostic material for deficiencies of minerals during pregnancy.

Amniotic fluid is necessary for the proper development of the embryo and fetus. It participates, among others, in nourishing and protecting the newly developing organism and performing information role in diagnostic procedures. The water contained in the amniotic fluid comes originally from maternal plasma and penetrates through the fetal membranes on the hydrostatic and osmotic way. As the placenta and fetal vessels develop, water and substances dissolved in maternal plasma pass through the placenta to the fetus and then into the amniotic fluid. In the period from 10 to 20 weeks of pregnancy, the composition of amniotic fluid is similar to that of fetal plasma. During this time, rapid bilateral diffusion between the fetus and amniotic fluid is observed through the non-keratinized fetal skin and amniotic surfaces, placenta and umbilical cord, which are easily permeable to water and substances dissolved in it. The composition of the amniotic fluid depends largely on the mother's nutritional status and on the exposure of her body to toxic substances. The role of minerals contained in the amniotic fluid is not clear. Due to the fact that the fetus swallows amniotic fluid, it may be a significant nutrient source for him. For this reason, it is suggested that the content of elements in the amniotic fluid may be a valuable marker of the nutritional status of the fetus and its exposure to toxic compounds.

In summary, the relationship between the concentration of minerals contained in amniotic fluid, mother's blood serum and hair with the development of the fetus and the occurrence of diseases complicating pregnancy requires further analysis. Planned research can significantly contribute to expanding knowledge in this topic. Based on the extremely important role of minerals in the normal functioning of the body of an adult human, it is particularly reasonable to conduct research to determine their significance at the stage of fetal life.

Research goals:

1. Prospective determination of the concentration of selected, essential and toxic elements in the blood serum of women in the second trimester of pregnancy.
2. Prospective determination of the concentration of selected, essential and toxic elements in the amniotic fluid.
3. Prospective determination of the concentration of selected, essential and toxic elements in hair taken from women in the second trimester of pregnancy.
4. Determination of the correlation between mineral components in the amniotic fluid, hair and mother's serum and parameters of fetal development and the state of health of the newborn.
5. Prospective determination of the diet of pregnant women, with particular emphasis on the supply of minerals.
6. Determination of the correlation between the diet of pregnant women and the concentration of selected minerals in amniotic fluid, mother's blood serum and hair.

Research assumptions:

Material for prospective studies will be collected during standard diagnostic procedures for patients at the gynecology and obstetrics clinic.

On the day of inclusion in the study, the patient will be collected blood from the ulnar vein - 5ml as part of a routine prenatal visit.

The following will be marked in the blood serum:

* concentration of minerals,
* placental capacity markers (pregnancy associated plasma protein A (PAPP-A), human chorionic gonadotropin (HCG), alfa-fetoprotein (AFP)).

The hair sample (about 0.5 g) from pregnant women will be taken on the day of inclusion in the study.

The pregnant women will be asked to complete a 3-day nutritional interview and nutritional survey.

From patients qualified for invasive prenatal diagnosis (amniocentesis), a sample of amniotic fluid (5 ml) will be taken, in which, in addition to the standardly evaluated parameters, selected mineral components will be marked.

Amniotic fluid samples will be collected during the routine amniocentesis procedure in patients with prenatal indications in 15-30 weeks of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed intrauterine pregnancy until week 14.
2. Single pregnancy without congenital malformations in ultrasound examination.
3. Lack of exponents threatening miscarriage (bleeding, lower abdominal pain, chorionic hematoma).
4. Lack of use of drugs affecting the mineral metabolism of the body.
5. Signing consent to participate in the study.

Exclusion Criteria:

1. Ectopic or heterotopic pregnancy.
2. Twin pregnancy (or other multiple pregnancy).
3. Obstetric load in the direction of numerous miscarriages, premature births under 34 weeks, pregnancy, fetal growth disorders (hypotrophy, macrosomia).
4. Congenital and /or genetic defects found in current pregnancy or in the patient.
5. Supply of drugs affecting the mineral metabolism of the body.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: A group of approximately 300 women is planned to be included in the study in the first trimester of pregnancy (up to 14 weeks of pregnancy).
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
minerals (Ca, Mg, Fe, Zn) | 1 year
  measure minerals in serum, hair, amniotic fluid

SECONDARY OUTCOMES:
maternal anthropometric parameters | 2 years
  measure weight in kilograms
fetal body weight | 2 years
  measure body weight according to ultrasound
fetal head circumference | 2 years
  measure head circumference according to ultrasound procedures
fetal biparietal diameter | 2 years
  measure biparietal diameter according to ultrasound procedures
prenatal diagnosis: PAPP-A | 2 years
  measure PAPP-A in maternal serum
prenatal diagnosis: HCG | 2 years
  measure HCG in maternal serum
prenatal diagnosis: AFP | 2 years
  measure AFP in maternal serum
dietary intake | 2 years
  measure energy, fat, proteins, carbohydrates and minerals intake

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland